CLINICAL TRIAL: NCT04504734
Title: Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study of Bucillamine in Patients With Mild-Moderate COVID-19
Brief Title: Bucillamine in Treatment of Patients With COVID-19
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Met definition of futility according to DSMB
Sponsor: Revive Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RT-003
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — bucillamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Bucillamine low dose (Active Comparator): Bucillamine 100 mg 3 times a day (TID)
  Interventions: Drug: Bucillamine
- Bucillamine high dose (Active Comparator): Bucillamine 200 mg 3 times a day (TID)
  Interventions: Drug: Bucillamine
- Placebo (Placebo Comparator): Placebo, 3 times a day (TID)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bucillamine — 100mg tablets
  Arms: Bucillamine low dose
Drug: Placebo — 100mg tablets
  Arms: Placebo
Drug: Bucillamine — 200mg tablets
  Arms: Bucillamine high dose

SUMMARY:
This is a Phase 3, multi-center, randomized, double blind, placebo controlled, clinical study of bucillamine (2 dosage levels) in patients with mild-moderate COVID-19. Patients will be randomized 1:1:1 to receive bucillamine 100 mg 3 times a day (TID), bucillamine 200 mg TID or placebo TID for up to 14 days. After the first interim analysis when a single dose is selected, patients will then be randomized 1:1 to the selected bucillamine dose or placebo. This dose has now been chosen as 600 mg. The study will be overseen by an independent Data and Safety Monitoring Board (DSMB). Up to 50 centers in the United States will conduct this study. Up to 1000 patients will be enrolled in this study. Patients will participate in the study approximately 45 days.

DETAILED DESCRIPTION:
This is a Phase 3, multi-center, randomized, double blind, placebo controlled, clinical study of bucillamine (2 dosage levels) in patients with mild-moderate COVID-19. Patients will be randomized 1:1:1 to receive bucillamine 100 mg 3 times a day (TID), bucillamine 200 mg TID or placebo TID for up to 14 days. After the first interim analysis when a single dose is selected, patients will then be randomized 1:1 to the selected bucillamine dose or placebo. This dose has now been chosen as 600 mg. The study will be overseen by an independent Data and Safety Monitoring Board (DSMB). Up to 50 centers in the United States will conduct this study.

Patients qualifying for study enrollment will initiate therapy as outpatients, under home quarantine. Patients will receive continued standard care of therapy (per study site written policies or guidelines) together with bucillamine and/ or matching placebo for up to 14 days. Dosing should continue until the treatment course is completed or as medically indicated (e.g., deterioration of clinical status and alternative therapy required). If the patient requires hospitalization during the study period, treatment will be discontinued.

Following completion of the treatment course, follow up assessments will be performed by a study nurse 14, 28, 42, and 60 days following the end of treatment.

Up to 1000 patients will be enrolled in this study. Patients will participate in the study approximately 45 days.

ELIGIBILITY:
Inclusion Criteria:

* Is within 72 hours from onset of symptoms consistent with COVID 19 at time of study enrollment
* Has at least 2 of the following: fever (oral temperature ≥38°C), cough, shortness of breath, chest x ray changes consistent with COVID-19 at time of screening
* Has peripheral capillary oxygen saturation (SpO2) ≥94 by pulse oximetry at time of screening
* Has either a laboratory-confirmed SARS-CoV-2 infection as determined by FDA-approved rapid diagnostic (e.g., PCR) assay
* Has a score of ≤ 2 on the 8-category NIAID ordinal scale at time of screening
* Agrees to the collection of blood and urine samples, nasopharyngeal (NP) swabs, and non-invasive oxygen monitoring (via pulse oximeter) per protocol
* Patient (or their legally authorized representative) is willing and able to provide written informed consent prior to performing study procedures
* Understands and agrees to comply with planned study procedures
* Women of childbearing potential must agree to either abstinence or use at least 1 primary form of contraception not including hormonal contraception from the time of screening through Day 29 following randomization. All subjects of childbearing potential, including males with partners of childbearing potential, must use highly effective methods of birth control defined as those, alone or in combination, that result in a low failure rate (i.e., less than 1 percent per year) when used consistently and correctly. Abstinence is NOT an acceptable method of contraception UNLESS it is the subject's normal practice.

Exclusion Criteria:

* Prior history of, or considered to be at risk for, agranulocytosis, nephropathy, liver disease, or interstitial pneumonia
* Serious hepatic disorder (Child-Pugh scores B or C) or alanine transaminase (ALT) or aspartate transaminase (AST) > 5 times the upper limit of normal (ULN) at screening
* Chronic kidney disease (CKD) National Kidney Foundation (NKF) stages 3B - 5 chronic renal dysfunction (estimated glomerular filtration rate [eGFR] <45 mL/min/1.73m2 according to Cockcroft Gault formula)
* Proteinuria ≥ 1+ or ≥ 30 mg on dipstick urinalysis that is confirmed on repeat assessment within 24 hours
* Serum BUN ≥ 2 × ULN or Cr ≥ 2 × ULN
* Leukopenia with absolute granulocyte count < 1500/µL
* History of positive Human Immunodeficiency virus (HIV) test or organ transplant
* Receipt of cancer chemotherapy or immunomodulatory drugs including (but not limited to) biologics such as anti-CD20, anti-TNF, anti-IL6; alkylating agents (e.g., cyclophosphamide); antimetabolites (e.g., azathioprine); or chronic corticosteroid use equivalent to prednisone >10 gm/day, during preceding 2 months
* Confirmed positive for influenza at screening
* Confirmed positive for respiratory syncytial virus (RSV) at screening
* Pregnant or breastfeeding
* Current use of, or known allergy to bucillamine or penicillamine (e.g., for Wilson's disease, rheumatoid arthritis)
* Current participation in any other clinical trial of an experimental treatment
* Receipt of any experimental treatment for COVID-19 (herbal/homeopathic, off-label, compassionate use, or trial related) within the 30 days prior to screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 713 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Efficacy: Frequency of hospitalization or death | From time of first dose through Day 28 following randomization
  Proportion of patients meeting a composite endpoint of hospitalization or death

SECONDARY OUTCOMES:
Safety: Changes in adverse events from baseline to end of study | From time of first dose through Day 28 following randomization
  Number of adverse events

CONTACTS AND LOCATIONS:
Locations (47):
- United States (46):
  - Cullman Clinical Trials, Cullman, Alabama
  - Avant Research Associates, LLC, Huntsville, Alabama
  - West Valley Research Clinic, Phoenix, Arizona
  - HealthStar Research LLC, Hot Springs, Arkansas
  - ASCADA Research, Huntington Beach, California
  - Samuel Ross MD Inc., Los Angeles, California
  - Amicis Research Center, Northridge, California
  - Optimus Medical Group, San Francisco, California
  - C & R Research Services USA, Coral Gables, Florida
  - Sweet Hope Research Specialty Inc, Hialeah, Florida
  - Encore Medical Research, Hollywood, Florida
  - Entrust Clinical Research, Kendall, Florida
  - Columbus Clinical Services, Miami, Florida
  - Verus Clinical Research, Miami, Florida
  - Nuren Medical & Research Center, Miami, Florida
  - Advance Medical Research Services Corp, Miami, Florida
  - Amavita Clinical Research, North Miami Beach, Florida
  - C & R Research Services USA, Tampa, Florida
  - Encore Medical Research of Weston LLC, Weston, Florida
  - Clinical Site Partners LLC, Winter Park, Florida
  - American Clinical Trials LLC, Acworth, Georgia
  - Quad Clinical Research LLC, Chicago, Illinois
  - Koch Family Medicine, Morton, Illinois
  - Revive Research Institute Inc., Farmington Hills, Michigan
  - SRI International, Plymouth, Michigan
  - Great Lakes Research Institute, Southfield, Michigan
  - Revival Research Institute LLC, Sterling, Michigan
  - Machuca Family Medicine, Las Vegas, Nevada
  - Prime Global Research, The Bronx, New York
  - OnSite Clinical Solutions, Charlotte, North Carolina
  - OnSite Clinical Solutions, LLC, Charlotte, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Superior Clinical Research, Smithfield, North Carolina
  - Superior Clinical Research, Yanceyville, North Carolina
  - Dayton Clinical Research, Dayton, Ohio
  - Pharmacorp Clinical Trials Inc., Charleston, South Carolina
  - Novaceut Clinical Research, Clarksville, Tennessee
  - Physicians Quality Care, Jackson, Tennessee
  - Inquest Clinical Research, Baytown, Texas
  - C & R Research Services USA, Houston, Texas
  - Encore Imaging and Medical Research, Houston, Texas
  - R & H Clinical Research Inc., Katy, Texas
  - FMC Science, Lampasas, Texas
  - Family Practice Center, McAllen, Texas
  - R & H Clinical Research Inc., Stafford, Texas
  - Renovatio Clinical, The Woodlands, Texas
- Dr. Orvil Martínez-Rivera, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided